CLINICAL TRIAL: NCT06750042
Title: Analysis of Motor Performance in Children with Duchene's Muscular Dystrophy
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor, Cairo University
Other Study IDs: analysis of motor performance
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Duchene's Muscular Dystrophy
Keywords: Duchene's muscular Dystrophy; Pulmonary Functions; Pediatrics; motor performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Duchene's muscular Dystrophy: age ranging from 6 to 16 years, diagnosed with Duchene's muscular Dystrophy (DMD) will participate in the study. They will be selected from the Pediatric Rehabilitation Center of Deraya University's outpatient clinic in El-Minia district, Minia-Egypt.

SUMMARY:
25 boys, ages ranging from 6 to 16 years, diagnosed with Duchene's muscular Dystrophy (DMD) will participated in the study. They will be selected from the Pediatric Rehabilitation Center of Deraya University's outpatient clinic in El-Minia district, Minia-Egypt. The outcome will be assessed motor performance will be assed by Bruininks-Oseretsky Test of Motor Proficiency Second Edition (BOT™-2) : balance, running speed and agility, bilateral coordination and strength and by Blue Cherry; Geratherm Respiratory. It is used to measure vital capacity (VC), forced expired volume in one second (FEV1), FEV1/FVC, FEV1/VC, and peak expiratory flow (PEF) to provide objective information for monitoring lung health.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis is Duchene's muscular Dystrophy only not other types,
* ambulated with or without assistance,
* oriented and endurance enough to understand orders to perform ventilation on the Blue Cherry; Geratherm Respiratory device.

Exclusion Criteria:

* any cognitive or neurological condition (other than Duchene's muscular Dystrophy),
* history of previous surgical operations that can affect pulmonary functions, and structural scoliosis

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 25 ages ranging from 6 to 16 years, diagnosed with Duchene's muscular Dystrophy will participate in this study. They were selected from Pediatric rehabilitation center of Deraya university out-patient clinic in El-Minia district, Minia,
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-12-27 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
motor performance | measured for one time
  motor performance will be assessed by Bruininks-Oseretsky Test of Motor Proficiency Second Edition (BOT™-2)
respiratory function | measured for only one time
  respiratory function by Blue Cherry; Geratherm Respiratory. It is used to measure respiratory function to provide objective information for monitoring lung health.

IPD SHARING:
Plan to Share IPD: Undecided